CLINICAL TRIAL: NCT00283114
Title: A Phase 1, Multi-Dose Study of SGN-33 (Anti-huCD33 mAb; HuM195; Lintuzumab) in Patients With Acute Myeloid Leukemia and Myelodysplastic Syndrome
Brief Title: A Safety Study of Lintuzumab in Patients With Acute Myeloid Leukemia and Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SG033-0001
Record Dates: First submitted 2006-01-25; First posted 2006-01-27 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome; Myeloproliferative Disorders; Chronic Myelomonocytic Leukemia
Keywords: Lintuzumab; Antigens, CD33; Antibodies, Monoclonal; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Hematologic Diseases; Myeloproliferative Disorders; Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Myeloproliferative Disorders; Leukemia, Myelomonocytic, Chronic; Hematologic Diseases; Leukemia | interventions — lintuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: lintuzumab

INTERVENTIONS:
Drug: lintuzumab — 1.5 - 8 mg/kg IV (in the vein) on Days 1, 8, 15, 22 and 29 of Cycle 1; 1.5 - 8 mg/kg IV (in the vein) every other week for all subsequent cycles
  Other Names: SGN-33

SUMMARY:
Phase 1a is an open-label, multi-dose, single-arm, dose-escalation study to define the toxicity profile, pharmacokinetics, and antitumor activity of SGN-33 in patients with myelodysplastic syndrome (MDS), acute myelogenous leukemia(AML), and CD33+ myeloproliferative diseases. Phase 1b includes patients with AML or MDS treated at the highest tolerated dose from phase 1a.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a diagnosis of MDS or AML.
2. Patients must have an ECOG performance status ≤ 2 and a life expectancy > 3 months.

Exclusion Criteria:

1. Patients who have received prior therapy with gemtuzumab ozogamicin (Mylotarg®) or other anti-CD33 monoclonal antibody treatment.
2. Patients with a prior allogeneic transplant.
3. Patients with known leptomeningeal or CNS involvement of leukemia. Patients with onset of CNS symptoms within the past 12 months will also be excluded.
4. Patients receiving chemotherapy within the last four weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2005-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
The incidence of adverse events and lab abnormalities. | 13 months
Pharmacokinetic (PK) profile and immunogenicity (Human Anti-Human Antibody; HAHA). | 13 months
Antitumor activity. | 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sievers, M.D., Study Director — Seagen Inc.
Locations (9):
- United States (9):
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Cancer Care Specialists of Central Illinois, Decatur, Illinois
  - Indiana Oncology-Hematology Consultants, Indianapolis, Indiana
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - St. Vincent's Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Cancer Center of the Carolinas, Greenville, South Carolina
  - Scott & White Memorial Hospital, Temple, Texas

REFERENCES:
- [Result] Raza A, Jurcic JG, Roboz GJ, Maris M, Stephenson JJ, Wood BL, Feldman EJ, Galili N, Grove LE, Drachman JG, Sievers EL. Complete remissions observed in acute myeloid leukemia following prolonged exposure to lintuzumab: a phase 1 trial. Leuk Lymphoma. 2009 Aug;50(8):1336-44. doi: 10.1080/10428190903050013. PMID 19557623